CLINICAL TRIAL: NCT03579784
Title: Biomarker-oriented Study of Durvalumab (MEDI4736) in Combination With Olaparib and Paclitaxel in Gastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Do-Youn Oh (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Do-Youn Oh, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-15-11655
Record Dates: First submitted 2018-06-19; First posted 2018-07-09 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — Paclitaxel; olaparib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab+Olaparib+Paclitaxel (Experimental): 1. st cycle : Paclitaxel+Olaparib
     * Olaparib 150mg bid on D1-28
     * Paclitaxel 80 mg/m2 mg iv on D1, D8, D15
  2. nd cycle and thereafter: Durvalumab+Olaparib+Paclitaxel :
     * Olaparib 150mg bid on D1-28
     * Durvalumab 1.5 g iv on D1
     * Paclitaxel 80 mg/m2 mg iv on D1, D8, D15 Every 4 weeks
  During first 4 weeks, palictaxel/olaparib dual combination will be used. Since 2nd cycle, palictaxel/olaparib/Durvalumab combination will be used.
  Interventions: Drug: Paclitaxel; Drug: Olaparib; Drug: Durvalumab

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 80 mg/m2 mg iv on D1, D8, D15 Every 4 weeks
Drug: Olaparib — Olaparib 150mg bid on D1-28 Every 4 weeks
Drug: Durvalumab — Durvalumab 1.5 g iv on D1 Every 4 weeks

SUMMARY:
<Research Hypothesis> The dynamics of immune systems by Olaparib and its changes by combination with immune-oncology agents will be uncovered.

The combination of Olaparib with Durvalumab with paclitaxel is tolerable and efficacious in gastric cancer.

<Objectives>

Primary Objectives:

To assess the effect of Durvalumab in combination with olaparib and paclitaxel on DCR (Disease control rate) in gastric cancer patients

-Disease control rate (based on RECIST v1.1)

Secondary Objective(s):

* Efficacy: overall response rate (RECIST 1.1, ir response), progression-free survival, duration of response, overall survival, overall survival at 6 month, overall survival at 1 year, EORTC QLQ-C30,
* Safety: toxicity (CTCAE V4.1), irAE

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age >= 19 years at time of study entry
3. Histologically proven gastric cancer
4. Unresectable or recurrent
5. Previous exposure to 1 palliative chemotherapy for their unresectable or recurrent cancer (Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing 5-Fluoropyrimidine monotherapy or 5-fluoropyrimidine and platinum based regimen is considered as first-line therapy)
6. Should have measurable lesion based on RECIST V1.1
7. Without previous expose to immune-oncology agents including anti-CTLA4, anti-PD1, anti-PDL1, etc
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 , and body weight >30 kg
9. Life expectancy of > 12weeks
10. Adequate normal organ and marrow function as defined below:

    * Haemoglobin ≥ 10.0 g/dL without transfusion within 28 days
    * No features of MDS/AML
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
    * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
    * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). <<This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>>
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
    * Serum creatinine CL>51 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
11. Female subjects must either be of non-reproductive potential or must have a negative serum pregnancy test upon study entry.

    Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
12. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)Previous enrollment or randomization in the present study
2. Participation in another clinical study with an investigational product during the last 3weeks
3. Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab
4. Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 28 days prior to the first dose of study drug (14 days prior to the first dose of study drug for subjects who have received prior TKIs [e.g., erlotinib, gefitinib and crizotinib] and within 6 weeks for nitrosourea or mitomycin C). (If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period may be required.)
5. Brain metastases or spinal cord compression unless the patient is stable (asymptomatic; no evidence of new or emerging brain metastases; and stable and off steroids for at least 14 days prior to start of study treatment). Following radiotherapy and/or surgery of the brain metastases subjects must wait 4 weeks following the intervention and before randomisation with imaging to confirm stability.
6. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction
7. Current or prior use of immunosuppressive medication within 14days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
8. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   -Subjects with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.

   Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
9. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Subjects with vitiligo or alopecia
    * Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Subjects without active disease in the last 5 years may be included but only after consultation with the study physician
    * Subjects with celiac disease controlled by diet alone
11. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
12. History of primary immunodeficiency
13. History of allogeneic organ transplant
14. History of hypersensitivity to durvalumab or any excipient
15. History of hypersensitivity to the combination or comparator agent
16. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
17. History of leptomeningeal carcinomatosis
18. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
19. Female subjects who are pregnant or breastfeeding or male or female subjects of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
20. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
21. Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
22. Subjects with uncontrolled seizures.
23. Features of MDS/ AML

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | 8weeks
  The percentage of patients who have achieved CR, PR, SD based on RECIST v1.1

SECONDARY OUTCOMES:
Overall response rate | 8weeks
  According to RECIST 1.1, ir response criteria
Progression-free survival | 8weeks
  Time from randomization until disease progression or death
Duration of response | 8weeks
  Time from documentation of tumor response to disease progression
Overall survival | 8weeks
  Time from randomization until death from any cause
Safety and tolerability as measured by number and grade of toxicity events | 2weeks
  Overall Safety Profile by CTCAE V4.1, irAE

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No